CLINICAL TRIAL: NCT03964350
Title: Behavior and Brain Responses to Drugs
Brief Title: Behavior Brain Responses
Acronym: BBR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB19-0293
Record Dates: First submitted 2019-05-15; First posted 2019-05-28 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Drinking; Drinking Behavior; Physiological Effects of Drugs; Central Nervous System Depression
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethanol (Experimental): Subjects will receive ethanol (0.4 or 0.8 g/kg) which will be administered in a gelatin vehicle.
  Interventions: Drug: Ethanol
- Placebo (gelatin vehicle) (Placebo Comparator): Subjects will receive placebo of black cherry sugar-free jello.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ethanol — The 0.8 g/kg body weight dose of gelatin alcohol will be divided into an average of 10 servings of 0.08 g/kg each. The 0.8 g/kg dose is equivalent to 4 standard drinks, where a standard drink is defined as one 12 oz beer, one 5 oz glass of wine, or one 1.5 oz shot of 80 proof alcohol.
  The 0.4 g/kg body weight dose of gelatin alcohol will be divided into an average of 5 servings of 0.08 g/kg each. The 0.4 g/kg dose is equivalent to 2 standard drinks, where a standard drink is defined as one 12 oz beer, one 5 oz glass of wine, or one 1.5 oz shot of 80 proof alcohol.
  Arms: Ethanol
Other: Placebo — The placebo comparator will be individual servings of back cheery sugar-free jello.
  Arms: Placebo (gelatin vehicle)

SUMMARY:
To compare responses to acute oral doses of ethanol in healthy young adults who experience mainly stimulant subjective effects from the drug or mainly sedative effects.

ELIGIBILITY:
* 21-35 years old
* 4-30 alcoholic drinks per week (as reported on PHQ or TLFB)
* No 'flushing' reaction to alcohol
* BMI 19-26
* High school education or greater, fluent in English
* No night shift work
* No current or past year Axis I psychiatric disorder including drug/alcohol dependence
* No current psychopharmacological treatment
* No lifetime ADHD or prescription for ADHD medication
* No abnormal EKG, cardiovascular illness, high blood pressure
* No medical condition or pharmacological treatment for which alcohol is contraindicated
* Not pregnant, lactating, or planning to become pregnant
* Smoke <6 cigarettes per day

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First (0 g/kg), Then Ethanol (0.4 g/kg), Then Ethanol (0.8 g/kg): Participants who received placebo first, then low dose ethanol then high dose ethanol
- Placebo (0 g/kg), Then Ethanol (0.8 g/kg), Then Ethanol (0.4 g/kg): participants who received placebo, then high dose ethanol then low dose ethanol
- Ethanol (0.4 g/kg), Then Ethanol (0.8 g/kg), Then Placebo (0 g/kg): participants who received low dose ethanol, then high dose ethanol, then placebo
- Ethanol First (0.8 g/kg) Then Ethanol (0.4 g/kg), Then Placebo (0 g/kg): Participants who received high dose ethanol first, then low dose ethanol, then placebo
- Ethanol First (0.8 g/kg), Then Placebo (0 g/kg), Then Ethanol (0.4 g/kg),: Participants who received high dose ethanol first, then placebo, then low dose ethanol
- Ethanol First (0.4 g/kg), Then Placebo (0 g/kg), Then Ethanol (0.8 g/kg),: Participants who received low dose ethanol first, then placebo, then high dose ethanol
Period: Overall Study
Arm/Group | Placebo First (0 g/kg), Then Ethanol (0.4 g/kg), Then Ethanol (0.8 g/kg) | Placebo (0 g/kg), Then Ethanol (0.8 g/kg), Then Ethanol (0.4 g/kg) | Ethanol (0.4 g/kg), Then Ethanol (0.8 g/kg), Then Placebo (0 g/kg) | Ethanol First (0.8 g/kg) Then Ethanol (0.4 g/kg), Then Placebo (0 g/kg) | Ethanol First (0.8 g/kg), Then Placebo (0 g/kg), Then Ethanol (0.4 g/kg), | Ethanol First (0.4 g/kg), Then Placebo (0 g/kg), Then Ethanol (0.8 g/kg),
Started | 6 | 5 | 3 | 6 | 6 | 4
Sedative-like Effects | 3 | 3 | 1 | 3 | 3 | 2
Stimulant Like Effects | 3 | 2 | 2 | 3 | 3 | 2
Completed | 6 | 5 | 3 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sedative-like Effects (All Study): Subjects that experienced more sedative like effects
- Stimulant-like (All Study): Subjects that experienced more stimulant-like effects
- Total: Total of all reporting groups
Arm/Group | Sedative-like Effects (All Study) | Stimulant-like (All Study) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Number; unit: years]
  >21 years of age | 15 | 15 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Education - High School Education [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Subscales of the Drug Effects Questionnaire Across Sessions
Description: Participants will complete The Drug Effects Questionnaire during the initial baseline session to determine their subjective alcohol profile. The Drug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states : "Feel Drug", "Feel High", "Like Drug", and "Want More". All sub-scales ("Feel Drug", "Feel High", "Like Drug", and "Want More") are scored on a visual analogue scale (scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: At expected peak drug effect (30 min post drink administration)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (Gelatin): Subjects gelatin vehicle.
- Ethanol (0.4 g/kg): Low dose ethanol
- Ethanol (0.8 g/kg): High dose ethanol
Arm/Group | Placebo (Gelatin) | Ethanol (0.4 g/kg) | Ethanol (0.8 g/kg)
Number analyzed (Participants) | 30 | 30 | 30
units on a scale
  "Feel Drug" | 3.65 (15.9) | 45.5 (24.9) | 62.3 (20.3)
  "Feel High" | 3.0 (15.9) | 33.7 (27.4) | 47.0 (32.8)
  "Like Drug" | 10.0 (19.7) | 48.3 (22.7) | 60.9 (22.8)
  "Want More" | 10.1 (23.6) | 39.6 (30.4) | 45.3 (31.2)
Statistical Analysis 1: Comparison: Placebo (Gelatin) vs Ethanol (0.4 g/kg) vs Ethanol (0.8 g/kg); Test type: Superiority; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks
Groups:
- Ethanol (0.4 g/kg): Subjects will receive ethanol (0.4 g/kg) which will be administered in a gelatin vehicle.
- Ethanol (0.8 g/kg): Subjects will receive ethanol (0.8 g/kg) which will be administered in a gelatin vehicle.
Arm/Group | Ethanol (0.4 g/kg) | Placebo (Gelatin Vehicle) | Ethanol (0.8 g/kg)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03964350/Prot_SAP_000.pdf